CLINICAL TRIAL: NCT00318708
Title: Asthma Clinical Research Network (ACRN) Trial - Macrolides in Asthma (MIA)
Acronym: MIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Distinguished Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 377; U10HL074231 (NIH); 5U10HL074231 (NIH); 7U10HL074206 (NIH); 5U10HL074208 (NIH); 5U10HL074073 (NIH); 5U10HL074227 (NIH); 5U10HL074225 (NIH); 5U10HL074204 (NIH); 5U10HL074218 (NIH); 5U10HL074212 (NIH)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Clarithromycin; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clarithromycin + fluticasone (Experimental): clarithromycin 500 mg twice daily (Biaxin) + fluticasone propionate 88 mcg twice daily (Flovent® HFA 44 mcg two puffs twice daily)
  Interventions: Drug: clarithromycin; Drug: fluticasone propionate
- placebo + fluticasone (Active Comparator): placebo clarithromycin twice daily + fluticasone propionate 88 mcg twice daily (Flovent® HFA 44 mcg two puffs twice daily)
  Interventions: Drug: fluticasone propionate; Drug: placebo clarithromycin

INTERVENTIONS:
Drug: clarithromycin — clarithromycin 500 mg twice daily (Biaxin)
  Other Names: Biaxin
  Arms: clarithromycin + fluticasone
Drug: fluticasone propionate — fluticasone propionate 88 mcg twice daily (Flovent® HFA 44 mcg two puffs twice daily)
  Other Names: Flovent®
Drug: placebo clarithromycin — placebo clarithromycin twice daily
  Other Names: placebo Biaxin
  Arms: placebo + fluticasone

SUMMARY:
Asthma can be caused by a variety of factors, including tobacco smoke, allergens, and respiratory airway infections. Many people use inhaled corticosteroid medications to treat their symptoms. These medications, however, are not effective for everyone. Clarithromycin is an antibiotic that may effectively treat asthma in these individuals. This study will evaluate the effectiveness of clarithromycin at controlling asthma symptoms.

DETAILED DESCRIPTION:
Asthma prevalence has steadily increased in the United States since the early 1980s; currently, more than 20 million people are diagnosed with asthma. Individuals with this disease may experience periodic attacks of wheezing, shortness of breath, chest tightness, and coughing. While there are many known causes of asthma, including tobacco smoke and other allergens, the exact cause of some asthma cases remains unknown. Research has shown that in some individuals, respiratory airway infections may play a role in the onset and severity of the disease. Inhaled corticosteroids are commonly used to treat asthma; however, they do not effectively control symptoms for everyone. Clarithromycin, an antibiotic medication used to treat bacterial infections, may be an effective asthma treatment for individuals who do not respond well to inhaled corticosteroids. The purpose of this study is to evaluate the effectiveness of clarithromycin at reducing asthma symptoms.

This study will begin with a 4-week run-in period to standardize participants' asthma medication usage. During this time, all participants will stop their current asthma medications and instead will receive inhaled fluticasone twice a day. Albuterol will be available as a rescue medication if necessary. Study visits will take place every 2 weeks. Blood and saliva samples will be obtained for laboratory tests and participants will complete standardized questionnaires to assess asthma symptoms and quality of life. Spirometry will be performed to measure lung function. Medication adherence will be monitored with a daily diary and an electronic pill counting device. At the end of Week 4, participants will be evaluated for study eligibility. If eligible, participants will undergo a bronchoscopy and a lung biopsy to test for Mycoplasma pneumoniae and Chlamydia pneumoniae, two bacteria that have been identified as possible factors in the development of asthma.

The treatment phase of the study will last 16 weeks. Participants will be randomly assigned to receive either 500 mg of clarithromycin or placebo twice a day, plus inhaled fluticasone. At monthly study visits, spirometry and blood collection will be performed. Standardized questionnaires to assess asthma symptoms will be completed every 2 weeks. Medical adherence will continue to be monitored. At the end of Week 16, participants will stop receiving clarithromycin or placebo, but will continue to receive fluticasone. Asthma symptoms, rescue medication usage, quality of life, and lung capacity will be assessed; tissue samples will be examined for the presence of Mycoplasma pneumoniae and Chlamydia pneumoniae. An 8-week washout period will follow to observe any lingering medication effects and to monitor for safety. Monthly study visits during this period will include spirometry and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* History of physician-diagnosed asthma
* Methacholine PC20 less than or equal to 16 mg/ml and/or FEV1 improvement greater than or equal to 12% in response to 180 mcg albuterol
* Stable asthma for at least 6 weeks prior to study entry
* FEV1 greater than or equal to 60% of predicted result following 180 mcg albuterol
* Juniper ACQ score greater than or equal to 1.5 (optimal ACQ score cut-off point for asthma that is "not well-controlled" by NIH/Global Initiative for Asthma [GINA] guidelines)
* Nonsmoker (less than 10 pack-per-year lifetime smoking history and no smoking in the year prior to study entry)
* Able to perform spirometry, as per American Thoracic Society criteria
* 75% adherence with diary cards, fluticasone (monitored with Doser), and placebo pill trial (monitored electronically with Electronic Drug Exposure Monitor [eDEM] pill dose counter) for the final 2 weeks of the four-week run-in period
* At Visit 1, in steroid-naïve participants, no significant adrenal suppression, defined as a plasma cortisol concentration less than 5 mcg/dL. If adrenal suppression occurs, a 250 mcg corticotropin (ACTH) stimulation test will be performed. Plasma cortisol levels will be collected at baseline, and 30 and 60 minutes after the ACTH stimulation test. Participants must have a cortisol concentration greater than 20 mcg/dL on at least one of the post-ACTH time points
* Absence of bronchoscopy-induced exacerbation; if bronchoscopy-induced exacerbation has occurred, prednisone therapy must have stopped at least 6 weeks prior to study entry
* Absence of respiratory tract infection; if infection has occurred, infection-related symptoms must have stopped at least 6 weeks prior to study entry
* Has experienced no more than two exacerbations or respiratory tract infections prior to study entry
* If female and able to conceive, willing to utilize two medically acceptable forms of contraception (one non-barrier method with single barrier method OR double barrier method)

Exclusion Criteria:

* Presence of lung disease other than asthma
* Presence of vocal cord dysfunction, due to potential confounding of ACQ score
* Significant medical illness other than asthma
* History of atrial or ventricular tachyarrhythmia
* Use of any medication that has a significant interaction with clarithromycin, including herbal or alternative therapies
* Asthma exacerbation within 6 weeks of the screening visit or during the run-in period prior to bronchoscopy
* Use of systemic steroids or change in dose of controller therapy within 6 weeks of the screening visit
* Inability, in the opinion of the study investigator, to coordinate use of dry powder or metered-dose inhaler or to comply with medication regimens
* Inability or unwillingness to perform required study procedures
* Prolonged heart rate corrected QT-interval (greater than 450 msec in women and greater than 430 msec in men) on echocardiogram (ECG) at study entry
* Low potassium or magnesium levels (based on local Asthma Clinical Research Network laboratory definitions)
* Abnormal elevation of liver function tests (AST, ALT, total bilirubin, or alkaline phosphatase)
* Abnormal prothrombin time (PT) or partial thromboplastin time (PTT) results
* Reduced creatinine clearance
* Contraindication to bronchoscopy, as determined by medical history or physical examination
* Regular consumption of grapefruit or grapefruit juice
* Pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Calhoun, MD, Principal Investigator — University of Texas, Galveston; Mario Castro, MD, Principal Investigator — Washington University School of Medicine; Robert F. Lemanske, MD, Principal Investigator — University of Wisconsin, Madison; Richard J. Martin, MD, Principal Investigator — National Jewish Health; Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital; Stephen P. Peters, MD, PhD, Principal Investigator — Wake Forest University Health Sciences; Homer A. Boushey, MD, Principal Investigator — University of California, San Francsico; Stephen I. Wasserman, MD, Principal Investigator — University of California, San Diego; Emily DiMango, MD, Principal Investigator — Columbia University; Monica Kraft, MD, Principal Investigator — Duke University; Reuben M Cherniack, MD, Study Chair — National Jewish Health
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin

REFERENCES:
- [Result] Sutherland ER, King TS, Icitovic N, Ameredes BT, Bleecker E, Boushey HA, Calhoun WJ, Castro M, Cherniack RM, Chinchilli VM, Craig TJ, Denlinger L, DiMango EA, Fahy JV, Israel E, Jarjour N, Kraft M, Lazarus SC, Lemanske RF Jr, Peters SP, Ramsdell J, Sorkness CA, Szefler SJ, Walter MJ, Wasserman SI, Wechsler ME, Chu HW, Martin RJ; National Heart, Lung and Blood Institute's Asthma Clinical Research Network. A trial of clarithromycin for the treatment of suboptimally controlled asthma. J Allergy Clin Immunol. 2010 Oct;126(4):747-53. doi: 10.1016/j.jaci.2010.07.024. PMID 20920764
- See also: Click here for the Asthma Clinical Research Network (ACRN) web site — http://www.acrn.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Fluticasone: placebo clarithromycin + fluticasone propionate 88 mcg twice daily (Flovent® HFA 44 mcg two puffs twice daily)
Period: Overall Study
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Started | 47 | 45
8-week Milestone | 42 | 42
Completed | 39 | 40
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Clarithromycin + Fluticasone: Clarithromycin 500 mg bid (Biaxin) + fluticasone propionate 88 mcg bid (Flovent® HFA 44 mcg two puffs bid)
- Placebo + Fluticasone: Fluticasone propionate 88 mcg bid (Flovent® HFA 44 mcg two puffs bid)
- Total: Total of all reporting groups
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 45 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.5) | 37.5 (10.5) | 39.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United States | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Juniper Asthma Control Questionnaire (ACQ) Results
Description: The Juniper asthma control questionnaire (ACQ) consists of six questions answered by the asthma patient with respect to symptoms, rescue medication use, and night-time awakenings due to asthma. A seventh item in the ACQ is the percent predicted FEV1. Each of the seven items is scored from from 0 (best) to 6 (worst), and then the seven items are averaged to yield a number from 0 (best) to 6 (worst). Asthma patients needed to display an ACQ greater than or equal to 1.25 in order to be eligible for randomization. A reduction of 0.5 units or more in the ACQ over the 16 weeks of treatment is considered to be clinically significant.
Time Frame: Measured every four weeks during the 16-week treatment period, with the change (week 16 minus baseline) as the primary outcome
Population: The number of participants for the analysis was determined as the number who completed the full 16 weeks (value at 16 weeks minus value at baseline).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
units on a scale | -0.15 (0.14) | -0.38 (0.14)

2. Secondary Outcome: Asthma Rescue Medication Use
Description: number of rescue puffs per day
Time Frame: the week-16 average minus the baseline-week average
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: rescue puffs per day
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
rescue puffs per day | -0.71 (0.23) | -0.14 (0.24)

3. Secondary Outcome: AM Peak Expiratory Flow (PEF)
Description: daily AM peak expiratory flow (PEF) measured in liters per minute
Time Frame: the week-16 average minus the baseline-week average
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters per minute
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
liters per minute | 8.31 (4.55) | 11.69 (4.48)

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: Forced expiratory volume in one second (FEV1) from spirometry
Time Frame: the week-16 value minus the baseline-value
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
Liters | -0.08 (0.05) | -0.06 (0.06)

5. Secondary Outcome: Methacholine Provocative Concentration (PC20)
Description: Logarithm-base 2 transformed Methacholine provocative concentration (PC20) based on FEV1
Time Frame: the week-16 value minus the baseline-value
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logarithm-base 2 of mg/mL
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
logarithm-base 2 of mg/mL | 1.39 (0.30) | 0.41 (0.30)

6. Secondary Outcome: Exhaled Nitric Oxide (eNO)
Description: Exhaled nitric oxide (eNO) measured in parts per billion
Time Frame: the week-16 value minus the baseline-value
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
parts per billion | -0.33 (3.16) | 3.04 (3.26)

7. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: The Asthma Quality of Life Questionnaire (AQLQ) consists of 32 questions, with each question ranging from 1 (worst) to 7 (best). The 32 questions are averaged to yield an overall score, which is reported here. Therefore, a positive change between the 16-week score and the baseline score represents improvement.
Time Frame: the week-16 value minus the baseline-value
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (1 through 7)
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Number analyzed (Participants) | 39 | 39
units on a scale (1 through 7) | 0.41 (0.16) | 0.59 (0.15)

ADVERSE EVENTS:
Time Frame: 6 months
Description: does not differ from clinicaltrials.gov definitions
Arm/Group | Clarithromycin + Fluticasone | Placebo + Fluticasone
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 9/47 | 7/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clarithromycin + Fluticasone (N=47) | Placebo + Fluticasone (N=45)
respiratory infections (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
gastrointestinal events (Gastrointestinal disorders) | 7 (9) | 3 (5)

LIMITATIONS AND CAVEATS:
Participants underwent endobronchial biopsy for characterization of lower airway status for M pneumoniae or C pneumoniae. The target sample size was 72 positives and 72 negatives. Only 80 and 12 were recruited, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No